CLINICAL TRIAL: NCT03537456
Title: A Multicentre, Open-label, Interventional, Pilot Trial to Assess the Performance and Tolerance of mRDX-02-17 Dermal Filler in the Facial Rejuvenation
Brief Title: Pilot Trial to Assess the Performance and Tolerance of mRDX-02-17 Dermal Filler in the Facial Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mesoestetic Pharma Group S.L. (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPMES/0118/MD
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Facial Rejuvenation
Keywords: Dermal Filler; Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: mRDX-02-17 is recommended for correction and treatment of wrinkles and dermal depressions, when administered by intradermal injection.
  This is a multi-center, open-label, non-randomized, single-group clinical investigation in subjects aged 35-65 years old seeking facial rejuvenation.
  Because it is a medical device with an innovative composition and that it is a first-in-human investigation, we preferred an exploratory approach for the investigation design. The main objectives and clinical endpoints are the performance and the safety profile of the investigational device.
  The total study duration will be approximately 3 months or 90 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mRDX-02-17 (Experimental): mRDX-02-17 is a dermal filler recommended for correction and treatment of wrinkles and dermal depressions, which are administered by intradermal injections. It encourages repair and restructuring of skin tissue, reducing the signs of aging and has the following indications:
  * Hypotrophic tissues
  * Tissue hypotonicity
  * Crow's feet
  * Glogau III - IV
  * Fiztpatrick I - VI
  * WSRS (Wrinkle Severity Ranking Scale): 2-5
  Interventions: Device: mRDX-02-17

INTERVENTIONS:
Device: mRDX-02-17 — mRDX -02-17 is a dermal filler recommended for the correction and treatment of wrinkles and dermal depressions.
  It is a sterile and viscous aqueous solution of hyaluronic acid in a concentration of 1.5% (p/v) with acetyl tetrapeptide-9 and palmitoyl tripeptide-5, as auxiliary ingredients which is administrated by intradermal injections.
  This medical device encourages repair and restructuring of skin tissue and reduces the signs of aging.
  mRDX -02-17 is indicated for patients with hypotrophic tissues, Crow's feet, Glogau III-IV, all skin photo types (Fitzpatrick I - VI) and a WSRS score (Wrinkle Severity Ranking Scale) from 2 to 5.

SUMMARY:
mRDX-02-17 is a device for facial beauty care composed of hyaluronic acid in a concentration of 1.5% (p/v), as a functional ingredient, recommended for the correction and treatment of wrinkles and dermal depressions.

The primary hypothesis of this clinical investigation is that, at 30 days after the 60 days of treatment with mRDX-02-17, the mean WSRS score assessed by the investigator will decrease with at least 0.5 points compared to baseline evaluation.

DETAILED DESCRIPTION:
Minimally invasive procedures (injectable dermal fillers) are among the techniques preferred by an increasing number of specialists in Aesthetics due to their clinical performance regarding volume restoration and favorable safety profile.

An evaluation of pre-clinical data was performed before the clinical investigation design.

Similar dermal fillers have been used in several clinical investigations in humans with a good rate of clinical success and good safety profiles.

During January - March 2018, review of the scientific literature was performed, to find similar investigations to determine the minimal clinically significant difference between Baseline and a period of 30 days after the end the treatment.

Considering the exploratory nature of this study and the fact that this investigation is first-in-human, the clinical investigation is designed to have a number of 7 study visits and a treatment period of 60 days.

In a similar dermal filler study, Takanobu Mashiko et al used a 5-grade WSRS and showed that at 4 weeks after treatment, they achieved a 1.7 ± 0.5 (mean ± SD) improvement between those visits.

The primary objectives included in the present clinical investigation are the performance of the medical device in terms of absolute change of Wrinkle Severity Rating Scale (WSRS) score assessed by Investigator at 90 days after the initiation of treatment with mRDX-02-17 dermal filler, compared to Baseline Visit (day 0), and overall safety of the medical device.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with age > 35 and ≤ 65 years;
* Subjects seeking tissue augmentation treatment on the face;
* Subjects willing to receive HA Filler for one and/or more mimetic and/or superficial facial wrinkles located in the facial area including periocular area;
* Subjects willing to receive HA Filler for one and/or more mimetic and/or superficial facial wrinkles;
* Subjects willing to provide signed informed consent to clinical investigation participation.

Exclusion Criteria:

* Use of aspirin and antiplatelet agents a week prior to treatment;
* Pregnant or lactating women;
* Subjects with a history of allergy or hypersensitivity to the HA or to other ingredients of the dermal filler;
* Subjects with hypersensitivity to salicylic acid or any of its derivates;
* Subjects with any dermal systemic pathologies, such as systemic lupus erythematosus, psoriasis, scleroderma etc.;
* Subjects presenting bleeding disorders in the past or present;
* Subjects taking or having indications for anticoagulant therapy;
* Use of concomitant treatments or procedures aimed to improve skin rejuvenation over the last six months before the clinical investigation enrolment, such as chemical peeling, dermabrasion, laser resurfacing;
* Subjects suffering from infectious diseases including herpes simplex virus infection, active hepatitis or human immunodeficiency virus;
* Subjects suffering from eczema, acne, and keloids;
* Subjects with any cutaneous manifested infection, disease or alteration;
* Subjects at risk in term of precautions, warnings, and contra-indications referred in the package insert of the clinical investigation device;
* Subjects with any facial aesthetic surgery in the preceding 12 months before the clinical investigation enrolment;
* Subjects with any active irritation or inflammation in the target areas of injection;
* Subjects who received botulinum toxin A injections in the face in the preceding 6 months;
* Subjects unlikely to cooperate in the clinical investigation or to comply with the treatment or with the clinical investigation visits;
* Subjects with solar activity, such as prolonged exposure to the sun, UV rays and extreme conditions of heat for at least a week after the treatment
* Direct or indirect contact with quaternary ammonium salts during the investigation
* Subjects participating in another clinical investigation or treated with another HA filler with the same indications at the same time or within the preceding 30 days.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-24 (Actual)

PRIMARY OUTCOMES:
Wrinkle Severity Rating Scale (WSRS) Score | 90 days
  The Wrinkle Severity Rating Scale is a 5-grade score scale, evaluating the severity of the facial wrinkles and comprising descriptive answers, numbered from 1 to 5. The best possible answer is 1 (no folds, continuos skin line) and the worst possible answer is 5 (extremely deep and long folds). This scale is evaluated by an investigator

SECONDARY OUTCOMES:
Wrinkle Severity Rating Scale (WSRS) Score | 0, 15, 30, 45, 60 and 90 days
  The Wrinkle Severity Rating Scale is a 5-grade score scale, evaluating the severity of the facial wrinkles and comprising descriptive answers, numbered from 1 to 5. The best possible answer is 1 (no folds, continuos skin line) and the worst possible answer is 5 (extremely deep and long folds). This scale is evaluated by the subject.
Global Aesthetic Improvement Scale (GAIS) Score | 15, 30, 45, 60 and 90 days
  The Global Aesthetic Improvement Scale is a 5-grade score scale, evaluating the general appearance, comprising descriptive answers, numbered from 1 to 5. The best possible answer is 1 (optimal cosmetic result) and the worst possible answer is 5 (the appearance is worse than the original condition). This scale is evaluated by the subject.
Treatment Satisfaction | 30 and 90 days
  Questionnaire related to Treatment satisfaction assessed by the subject
Choice of Recommendation | 90 days
  The choice of recommending further the treatment will be assessed by the subject at the final visit. It includes a 3-point scale. The subject must evaluate the treatment from the perspective of recommending it further by marking one of the the following answers: yes, perhaps or no.

OTHER OUTCOMES:
Number of adverse events | 0, 15, 30, 45, 60 and 90 days
  Collection of adverse events during each visit

CONTACTS AND LOCATIONS:
Overall Officials: Luis Luis, MD, Study Director — Medical Affairs Director
Locations (2):
- Romania (2):
  - Societatea Civila Medicala Doctor Rosu, Timișoara
  - Hyperclinica Medlife Sucursala Timisoara, Timișoara

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fitzgerald R, Graivier MH, Kane M, Lorenc ZP, Vleggaar D, Werschler WP, Kenkel JM. Update on facial aging. Aesthet Surg J. 2010 Jul-Aug;30 Suppl:11S-24S. doi: 10.1177/1090820X10378696. PMID 20844296
- [Background] Sudha PN, Rose MH. Beneficial effects of hyaluronic acid. Adv Food Nutr Res. 2014;72:137-176. doi: 10.1016/B978-0-12-800269-8.00009-9. PMID 25081082
- [Background] The European Medical Device Regulations Annex VIII. Classification rules. April 2017.
- [Background] ISO 14155:2011. Clinical investigation of medical devices for human subjects - Good clinical practice.
- [Background] Mashiko T, Kinoshita K, Kanayama K, Feng J, Yoshimura K. Perpendicular Strut Injection of Hyaluronic Acid Filler for Deep Wrinkles. Plast Reconstr Surg Glob Open. 2015 Dec 9;3(11):e567. doi: 10.1097/GOX.0000000000000552. eCollection 2015 Nov. PMID 26893992
- [Background] Kim BW, Moon IJ, Yun WJ, Chung BY, Kim SD, Lee GY, Chang SE. A Randomized, Evaluator-Blinded, Split-Face Comparison Study of the Efficacy and Safety of a Novel Mannitol Containing Monophasic Hyaluronic Acid Dermal Filler for the Treatment of Moderate to Severe Nasolabial Folds. Ann Dermatol. 2016 Jun;28(3):297-303. doi: 10.5021/ad.2016.28.3.297. Epub 2016 May 25. PMID 27274627
- [Background] Kopera D, Palatin M, Bartsch R, Bartsch K, O'Rourke M, Holler S, Baumgartner RR, Prinz M. An open-label uncontrolled, multicenter study for the evaluation of the efficacy and safety of the dermal filler Princess VOLUME in the treatment of nasolabial folds. Biomed Res Int. 2015;2015:195328. doi: 10.1155/2015/195328. Epub 2015 Mar 3. PMID 25821787
- [Background] Few J, Cox SE, Paradkar-Mitragotri D, Murphy DK. A Multicenter, Single-Blind Randomized, Controlled Study of a Volumizing Hyaluronic Acid Filler for Midface Volume Deficit: Patient-Reported Outcomes at 2 Years. Aesthet Surg J. 2015 Jul;35(5):589-99. doi: 10.1093/asj/sjv050. Epub 2015 May 11. PMID 25964628
- [Background] Callan P, Goodman GJ, Carlisle I, Liew S, Muzikants P, Scamp T, Halstead MB, Rogers JD. Efficacy and safety of a hyaluronic acid filler in subjects treated for correction of midface volume deficiency: a 24 month study. Clin Cosmet Investig Dermatol. 2013 Mar 20;6:81-9. doi: 10.2147/CCID.S40581. Print 2013. PMID 23687448
- [Background] Dong J, Gantz M, Goldenberg G. Efficacy and safety of new dermal fillers. Cutis. 2016 Nov;98(5):309-313. PMID 28040813
- [Background] De Boulle K, Heydenrych I. Patient factors influencing dermal filler complications: prevention, assessment, and treatment. Clin Cosmet Investig Dermatol. 2015 Apr 15;8:205-14. doi: 10.2147/CCID.S80446. eCollection 2015. PMID 25926750
- [Background] Rivkin AZ. Volume correction in the aging hand: role of dermal fillers. Clin Cosmet Investig Dermatol. 2016 Aug 30;9:225-32. doi: 10.2147/CCID.S92853. eCollection 2016. PMID 27621659
- [Background] Kuhne U, Esmann J, von Heimburg D, Imhof M, Weissenberger P, Sattler G. Safety and performance of cohesive polydensified matrix hyaluronic acid fillers with lidocaine in the clinical setting - an open-label, multicenter study. Clin Cosmet Investig Dermatol. 2016 Oct 20;9:373-381. doi: 10.2147/CCID.S115256. eCollection 2016. PMID 27799807
- [Background] Lorenc ZP, Bank D, Kane M, Lin X, Smith S. Validation of a four-point photographic scale for the assessment of midface volume loss and/or contour deficiency. Plast Reconstr Surg. 2012 Dec;130(6):1330-1336. doi: 10.1097/PRS.0b013e31826d9fa6. PMID 23190816
- [Background] Chen WY, Abatangelo G. Functions of hyaluronan in wound repair. Wound Repair Regen. 1999 Mar-Apr;7(2):79-89. doi: 10.1046/j.1524-475x.1999.00079.x. PMID 10231509
- [Background] McCall-Perez F, Stephens TJ, Herndon JH Jr. Efficacy and tolerability of a facial serum for fine lines, wrinkles, and photodamaged skin. J Clin Aesthet Dermatol. 2011 Jul;4(7):51-4. PMID 21779421
- [Background] Rzany B, Cartier H, Kestemont P, Trevidic P, Sattler G, Kerrouche N, Dhuin JC, Ma YM. Full-face rejuvenation using a range of hyaluronic acid fillers: efficacy, safety, and patient satisfaction over 6 months. Dermatol Surg. 2012 Jul;38(7 Pt 2):1153-61. doi: 10.1111/j.1524-4725.2012.02470.x. PMID 22759252
- [Background] Van Dyke S, Hays GP, Caglia AE, Caglia M. Severe Acute Local Reactions to a Hyaluronic Acid-derived Dermal Filler. J Clin Aesthet Dermatol. 2010 May;3(5):32-5. PMID 20725567
- [Background] Funt D, Pavicic T. Dermal fillers in aesthetics: an overview of adverse events and treatment approaches. Plast Surg Nurs. 2015 Jan-Mar;35(1):13-32. doi: 10.1097/PSN.0000000000000087. PMID 25730536
- [Background] Almeida A, Sampaio G. Hyaluronic acid in the rejuvenation of the upper third of the face: review and update - Part 1. 2018.
- [Background] Freedberg et al. Fitzpatrick's Dermatology In General Medicine (Two Vol. Set) 6th edition (May 23, 2003)
- [Background] ISO 14971:2012 Medical devices. Application of risk management to medical devices.
- [Background] ISO 13485:2016. Medical device - Quality management system- Requirements for regulatory purposes.
- [Background] ISO 10993: 2009. Part1. Biological evaluation of medical devices.
- [Background] ISO 14644: 2015 Part 1. Clean rooms and associated controlled environments.
- [Background] ISO 17665-1:2006. Sterilization of health care products -- Moist heat -- Part 1: Requirements for the development, validation and routine control of a sterilization process for medical devices
- [Background] Bhatt A. Protocol deviation and violation. Perspect Clin Res. 2012 Jul;3(3):117. doi: 10.4103/2229-3485.100663. No abstract available. PMID 23125964
- [Background] Ghooi RB, Bhosale N, Wadhwani R, Divate P, Divate U. Assessment and classification of protocol deviations. Perspect Clin Res. 2016 Jul-Sep;7(3):132-6. doi: 10.4103/2229-3485.184817. PMID 27453830
- [Background] MEDDEV 2.7/3 revision 3 Clinical Investigations: Serious Adverse Event Reporting Under Directives 90/385/EEC and 93/42/EEC.
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714